CLINICAL TRIAL: NCT03759548
Title: Nutritional Status and Pharmacological Treatment: Impact on the Toxicity and Quality of Life of Patients With Colorectal and Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Federal University of Minas Gerais (Other)
Collaborators: Mater Dei Hospital, Brazil (Other)
Responsible Party: Principal Investigator, Maria Isabel Toulson Davisson Correia, Clinical Professor, Federal University of Minas Gerais
Other Study IDs: CAAE: 91570318.5.0000.5149
Record Dates: First submitted 2018-11-15; First posted 2018-11-30 (Actual); Last update posted 2018-11-30 (Actual); Status verified 2018-11

CONDITIONS: Nutritional Status; Colorectal Cancer; Breast Cancer
Keywords: Nutritional Status; Colorectal Cancer; Breast Cancer; Pharmacological Treatment; Toxicity; Quality of Life
MeSH Terms: conditions — Colorectal Neoplasms; Breast Neoplasms | interventions — Nutrition Assessment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Breast Cancer: Breast Cancer's patients undergoing pharmacological treatments prior or after surgery.
  Interventions: Other: Assessment of nutritional status
- Colorectal Cancer: Colorectal Cancer's patients undergoing pharmacological treatments prior or after surgery.
  Interventions: Other: Assessment of nutritional status

INTERVENTIONS:
Other: Assessment of nutritional status — Observational study. Assessment of nutritional status.

SUMMARY:
Cancer patients undergo many different modalities of treatments. Pharmacological treatment should be well understood. The nutritional status is not taken into account when calculating drug's doses and this may have an impact in toxicity and quality of life. The present study proposes to evaluate the relationship between the calculation of pharmacological treatment's doses, the toxicity and the impact on quality of life among colorectal and breast cancer's patients.

DETAILED DESCRIPTION:
Cancer patients undergo various treatment modalities depending on tumor type, location, disease staging, and overall clinical conditions. Pharmacological treatments and surgeries are fundamental therapeutic strategies in many cases and are part of the daily routine of integrated cancer treatment services. The calculation of pharmacological doses often takes into account the patient's body surface area (BSA) or only weight, without however assessing their nutritional status as such. The surgical procedure, on the other hand, may expose the patient to an inflammatory response secondary to the operative trauma that requires immediate reaction of the diseased organism for an adequate recovery. In this sense, the objective of the present study is to evaluate the relationship between the calculated medication's doses and the nutritional status of patients submitted topharmacological treatment with neoadjuvant or adjuvant intention: patients candidates for surgery. Different instruments will be used for nutritional assessment, as well as a questionnaire on quality of life, a specific criterion for evaluation of toxicities, laboratory tests and imaging. Patients will be observed for 1 year and the data collected will allow the analysis of possible side effects and the impact on quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Pathological diagnosis of Colorectal Cancer or Breast Cancer
* Must have Performance Status to undergo surgery and pharmacological treatment (Adjuvant or Neoadjuvant treatment)

Exclusion Criteria:

* Non-operable patients
* Pacientes with poor Performance Status Eastern Cooperative Oncology Group (PS ECOG) >2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Colorectal or Breast Cancer undergoing Neoadjuvant or Adjuvant pharmacological treatment.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Impact in Quality of Life during pharmacological treatments | 1 year
  Impact in Quality of Life as assessed by European Organization for Research Treatment of Cancer (EORTC) Quality of life questionnaire (QLQ-C30)

SECONDARY OUTCOMES:
Pharmacological treatment-related adverse events | 1 year
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Locations (1):
- Rede Mater Dei de Saúde - Hospital Integrado do Câncer, Belo Horizonte, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No
Individual-level informations will not be available in order to preserve patient's identity.